CLINICAL TRIAL: NCT05739695
Title: Multicenter, Open-label, Prospective Randomized Controlled Trial of Radial Endobronchial Ultrasonography and Virtual Bronchoscopy Navigation for the Peripheral Pulmonary Lesions
Brief Title: A Trial of Radial EBUS Versus VBN for the Peripheral Pulmonary Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ilya Sivokozov (Other)
Responsible Party: Sponsor-Investigator, Ilya Sivokozov, Head of Respiratory Endoscopy Department, Central TB Research Institute
Organization: Central TB Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VBN-REBUS
Record Dates: First submitted 2022-02-04; First posted 2023-02-22 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer; Tuberculosis; Pneumonia
Keywords: navigation bronchoscopy; virtual bronchoscopy navigation; radial endobronchial ultrasound; BAL; TBLB
MeSH Terms: conditions — Lung Neoplasms; Tuberculosis; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VBN (Experimental): Virtual bronchoscopy
  Interventions: Diagnostic Test: Virtual bronchoscopy navigation
- VBN+rEBUS (Experimental): Combination of VBN and radial EBUS
  Interventions: Diagnostic Test: Virtual bronchoscopy navigation; Diagnostic Test: radial EBUS
- rEBUS (Active Comparator): Radial EBUS as a gold standard
  Interventions: Diagnostic Test: radial EBUS

INTERVENTIONS:
Diagnostic Test: Virtual bronchoscopy navigation — It is planned to use VBN as the only navigation technique to compare it with rEBUS
  Arms: VBN; VBN+rEBUS
Diagnostic Test: radial EBUS — It is planned to use rEBUS as the only navigation technique to compare it with VBN
  Arms: VBN+rEBUS; rEBUS

SUMMARY:
Peripheral pulmonary lesions are of growing importance in respiratory field. Early detection of lung cancer, tuberculosis and other diseases often needs a bronchoscopic investigation with different types of navigation. Current randomized clinical study is intended to compare three different modalities of navigation in bronchial tree - virtual bronchoscopy (VBN), radial endobronchial ultrasound (EBUS) and combination of both techniques.

DETAILED DESCRIPTION:
Current randomized clinical study is intended to compare three different modalities of navigation in bronchial tree - virtual bronchoscopy, radial EBUS and combination of both techniques. Around 300 patients with incidentally detected peripheral pulmonary lesions will be enrolled in 9 centers among Russia. All patients after obtaining an informed consent will be randomized in 1:1:1 fashion to three study groups depending on type of navigation technique used. All patients will undergone navigational bronchoscopy with rEBUS (group A), VBN (group B) and rEBUS+VBN (group C), data on diagnostic efficacy and safety of each modality of navigation will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed unverified solitary or multiple (up to 3) peripheral pulmonary lesions (PPLs)
2. PPL size 5 - 40 mm
3. Actual chest CT scan (<31 days prior to navigation bronchoscopy), collimation 1 mm, pulmonary window, DICOM format
4. Age > 18 years
5. Signed Informed consent form
6. Willing and ability to undergone a navigational bronchoscopy

Exclusion Criteria:

1. Unability to undergone navigation bronchoscopy for any reason
2. Any malignant disease during last 36 months
3. Known central endobronchial lesion of any cause
4. HIV-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Efficacy of navigational bronchoscopy in each study arm | At the end of study enrollment
  Incidence of final diagnoses confirmed by navigational bronchoscopy for each study arm

SECONDARY OUTCOMES:
Efficacy of each endoscopic biopsy modality in confirmation of final diagnosis | At the end of study enrollment
  Incidence of final diagnoses confirmed by navigational bronchoscopy for bronchoalveolar lavage, brush and transbronchial lung biopsy separately

OTHER OUTCOMES:
Safety profile of each study arm | At the end of study enrollment
  Incidence of complications reported at each study arm procedures

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Sivokozov, MD PhD, Study Chair — Central TB Research Institute
Locations (6):
- Russia (6):
  - Chelyabinsk Regional Clinical Center of Oncology and Nuclear Medicine, Chelyabinsk
  - Kurgan Regional Oncological Dispensary, Kurgan
  - Central TB Research Institute, Moscow
  - P. Hertsen Moscow Oncology Research Institute, Moscow
  - National Medical Research Centre for Oncology, Rostov-on-Don
  - Tomsk Regional Oncological Dispensary, Tomsk

IPD SHARING:
Plan to Share IPD: No